CLINICAL TRIAL: NCT06236139
Title: Phase 1/2 Dose-Escalation and Cohort Study of STEAP1 CART With Enzalutamide in Participants With mCRPC
Brief Title: Cell Therapy (STEAP1 CART) With Enzalutamide for the Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: PromiCell Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RG1123855; NCI-2023-10316 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20204 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-01-09; First posted 2024-02-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Cyclophosphamide; enzalutamide; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (STEAP1 CART, enzalutamide) (Experimental): Patients undergo leukapheresis then receive cyclophosphamide IV and fludarabine IV on days -5, -4 and -3 and STEAP1 CART IV on day 0. Patients may receive enzalutamide PO on day 0 then QD in the absence of disease progression or unacceptable toxicity. Patients also undergo a tumor biopsy at baseline, day 14 and optionally at progression. Patients additionally undergo blood sample collection, NM bone scan and CT scan, or MRI or PET scan throughout study. Additionally, patients may undergo ECHO or MUGA at screening.
  Interventions: Biological: Anti-STEAP1 CAR T-cells; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Enzalutamide; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Anti-STEAP1 CAR T-cells — Given IV
  Other Names: Anti-STEAP1 CAR T Cells; Anti-STEAP1 CAR-T Cells; STEAP1 CAR-T Cells; STEAP1-targeting CAR T-cells
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo NM bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis; Leukocyte Adsorptive Apheresis; White Blood Cell Reduction Apheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning; RNV Scan
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I/II trial tests the safety and effectiveness of cell therapy (STEAP1 CART) with enzalutamide in treating patients with prostate cancer that continues to grow despite surgical or medical treatments to block androgen production (castration-resistant) and that has spread from where it first started (the prostate) to other places in the body (metastatic). Prostate cancer is the second leading cause of cancer deaths in men. Localized prostate cancer is often curable and even metastatic disease may respond to treatment for a few years. Despite multiple therapies, including hormone therapy and chemotherapy, metastatic castration-resistant prostate cancer (mCRPC) still remains an incurable disease. Recently, adoptive cellular immunotherapies have been developed to transfer immunogenic cells to the patient to produce an anti-tumor response. Chimeric antigen receptor T (CART)-cell therapy is a type of treatment in which a patient's T-cells (a type of immune cell) are changed in the laboratory so they will attack tumor cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's tumor cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Prostate stem cell antigen and prostate specific membrane antigen CAR T cell therapies have been shown to be safe and effective, but objective tumor responses remain rare. STEAP1 is an antigen that promotes cancer growth and spread and is found to be broadly expressed in mCRPC tissues. STEAP1 CART is CAR T cells that have been engineered with a STEAP1 antigen to better target prostate tumor cells. Enzalutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of cancer cells. Giving STEAP1 CART with enzalutamide may kill more tumor cells in patients with mCRPC.

DETAILED DESCRIPTION:
OUTLINE: This is a dose escalation study of STEAP1 CART in combination with enzalutamide followed by a dose expansion study.

Patients undergo leukapheresis then receive cyclophosphamide intravenously (IV) and fludarabine IV on days -5, -4 and -3 and STEAP1 CART IV on day 0. Patients may receive enzalutamide orally (PO) on day 0 then once daily (QD) in the absence of disease progression or unacceptable toxicity. Patients also undergo a tumor biopsy at baseline, day 14 and optionally at progression. Patients additionally undergo blood sample collection, nuclear medicine (NM) bone scan and computed tomography (CT) scan, or magnetic resonance imaging (MRI) or positron emission tomography (PET) scan throughout study. Additionally, patients may undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening.

After completion of study treatment, patients are followed up at 2, 3, 4, 5, 6, 9, and 12 months then every 6 months up to year 5 followed by yearly up to year 15.

ELIGIBILITY:
Inclusion Criteria:

* Tissue confirmation of prostate adenocarcinoma
* Measurable disease by RECIST 1.1 criteria or bone only metastases with measurable PSA ( ≥ 1 ng/mL)
* Must have progressed (at least 2 rising PSA levels with at least a 1-week interval and a minimum PSA of 1.0 ng/mL, progression per RECIST 1.1, or 2 or more new bone lesions by bone scan), after becoming castration-resistant
* Have received the following for metastatic prostate cancer:

  * At least two lines of treatment
  * At least two Food and Drug Administration (FDA)-approved therapies with at least one being a second generation androgen receptor signaling inhibitor (e.g., abiraterone, darolutamide, apalutamide, or enzalutamide)
  * All available targeted therapies for which they are eligible in the metastatic setting (e.g., PARP inhibitors for BRCA 1/2 and immune checkpoint inhibitor for MSI-H or TMB-H ≥ 10 mut/Mb)
* Castrate levels of testosterone (< 50 ng/dL) with or without the use of androgen deprivation therapy
* 18 years or older at the time of enrollment
* Capable of understanding and providing a written informed consent
* Fertile male participants and their female partners must be willing to use an effective contraceptive method before, during, and for at least 4 months after the STEAP1 CART cell infusion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants will be permitted to receive radiation therapy for palliative purposes throughout the study period, except during the 2-week period prior to undergoing leukapheresis
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or estimated creatinine clearance > 50 mL/min as calculated using the Cockcroft-Gault formula and not dialysis dependent
* Total bilirubin ≤ 1.5 x ULN. Participants with suspected Gilbert syndrome may be included if Total bilirubin (Bili) > 3 mg/dL but no other evidence of hepatic dysfunction
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN
* ≤ grade 1 dyspnea and oxygen saturation (SaO2) ≥ 92% on ambient air
* If pulmonary function tests (PFTs) are performed based on the clinical judgement of the treating physician, participants with forced expiratory volume in 1 second (FEVI) >= 50% of predicted and diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) of >= 40% of predicted will be eligible
* Participants >= 60 years of age are required to have left ventricular ejection fraction (LVEF) evaluation performed within 1 year prior to lymphodepletion chemotherapy. LVEF may be established with echocardiogram or MUGA scan, and left ejection fraction must be >= 35%. Cardiac evaluation for other participants is at the discretion of the treating physician
* Absolute neutrophil count (ANC) > 1500 cells/ mm^3
* Hemoglobin > 9 g/dL
* Platelets > 100,000 per mm^3

Exclusion Criteria:

* Expecting to conceive or father children for the duration of the trial through 4 months after T cell infusion
* Active autoimmune disease: Participants with active autoimmune disease requiring immunosuppressive therapy are excluded. Case by case exemptions are possible with approval by principal investigator (PI)
* Corticosteroid therapy at a dose equivalent of >15 mg of prednisone per day (or equivalent). Pulsed corticosteroid use for disease control is acceptable
* Concurrent use of other investigational anti-cancer agents except for androgen deprivation therapy
* Active uncontrolled infection: human immunodeficiency virus (HIV) positive participants on highly active antiretroviral therapy (HAART) with a CD4 count > 500 cells/mm^3 are considered controlled, as are individuals with a history of hepatitis C who have successfully completed antiviral therapy with an undetectable viral load, and those with hepatitis B who have hepatitis well controlled on medication
* Uncontrolled concurrent illness: Participants may not have uncontrolled or concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia that would limit compliance with study requirements
* Untreated brain metastases: Participants with small asymptomatic brain metastases ( < 1 cm) or those with brain metastases previously treated and controlled with surgery or radiotherapy will be considered for inclusion at discretion of principal investigator, so long as all other eligibility criteria are met
* Active treatment for prior immune related adverse event to any immunotherapy: Participants receiving ongoing treatment for prior serious immune-related adverse events are excluded, with exception of hormone supplementation or corticosteroid therapy at equivalent of > 15 mg prednisone (or equivalent) per day, unless otherwise approved by PI
* Significant underlying neurologic disease: Study participants must not have significant active underlying neurologic disease, unless approved by PI. Peripheral neuropathy related to diabetes or prior chemotherapy is acceptable
* Other medical, social, or psychiatric factor that interferes with medical appropriateness and/or ability to comply with study, as determined by the PI
* Known allergic reactions to any of the components of study treatments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher adverse events (AEs) (Phase I) | Up to 28 days post infusion
  Toxicity will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Incidence of AEs (Phase II) | Up to 28 days post infusion
  Toxicity will be graded according to NCI CTCAE v 5.0.
Response (Phase II) | Up to 1 year post infusion
  Response will be defined as best overall response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and/or Prostate Cancer Working Group 3 (PCWG3) criteria.
Prostate specific antigen (PSA) response | At baseline up to 1 year post infusion
  PSA responses, defined as >= 50% reductions in PSA from baseline at any point post baseline assessment will be calculated.
Time to response (TTR) | At time from study infusion to time of first documented response up to 1 year post infusion
  TTR will be assessed from the time of study infusion to time of first documented response (partial response [PR] or better).
Duration of response (DOR) | At time of first documented response to time of confirmed progression up to 1 year post infusion
  DOR will be assessed from the time of first documented response (PR or better) to time of confirmed disease progression.

SECONDARY OUTCOMES:
Progression free survival (PFS) | At time from initiation of protocol treatment to disease progression or death up to 1 year post infusion
  PFS will be estimated using the method of Kaplan and Meier with time zero being the time of first T cell infusion.
Overall survival (OS) | At time from initiation of protocol treatment to death of any cause up to 1 year post infusion
  OS will be estimated using the method of Kaplan and Meier with time zero being the time of first T cell infusion.
Frequency of participants that achieve an overall response rate (ORR, including complete and partial response) according to RECIST v.1.1 or PCWG3 | Anti-tumor response according to RECIST v1.1 or PCWG3 up to 1 year post infusion
  To measure how well the treatment succeeds in producing the desired effect.
Frequency of participants that achieve a stable disease (SD) according to RECIST v.1.1 or PCWG3 | Anti-tumor response according to RECIST v1.1 or PCWG3 up to 1 year post infusion
  To measure how well the treatment succeeds in producing the desired effect.
Frequency of participants that achieve a clinical benefit rate (ORR + SD) stable disease RECIST v.1.1 or PCWG3 | Anti-tumor response according to RECIST v1.1 or PCWG3 up to 1 year post infusion
  To measure how well the treatment succeeds in producing the desired effect.
ORR by immune RECIST | Up to 1 year post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Nadal Rios, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No